CLINICAL TRIAL: NCT02944201
Title: Beta Adrenergic Receptor Blockade as a Novel Therapy for Patients With Adenocarcinoma of the Prostate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Benjamin Gartrell, Assistant Professor of Oncology, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-6632
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: carvedilol; biomarkers; autonomic nerves
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carvedilol (Experimental): Carvedilol will be started at 6.25 mg by mouth twice daily. Patients will take carvedilol for 28 days prior to prostatectomy. They will be seen every 7 days and adjustments in the dose will be considered at those visits.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol will give twice daily until prostatectomy
  Other Names: Coreg

SUMMARY:
This will be a single arm, window of opportunity study in men with treatment-naïve prostate cancer who will proceed to prostatectomy. Men will be treated with carvedilol prior to undergoing prostatectomy.

DETAILED DESCRIPTION:
Preclinical research has demonstrated that autonomic nerve fibers in the prostate gland regulate prostate cancer development and dissemination. Studies in human prostate cancer specimens indicate that higher densities of autonomic nerve fibers are associated with poor clinical outcomes.

In this clinical trial the beta-blocker carvedilol will be given to men diagnosed with prostate cancer. Men will begin carvedilol following their diagnostic prostate biopsy and will continue carvedilol until prostatectomy. The primary outcome measure is the change in Ki-67 and TUNEL assay biomarkers in prostate biopsy and prostatectomy tissues.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be able to provide study-specific informed consent prior to study entry.
2. Age ≥ 18
3. ECOG Performance Status 0-1
4. Pathologically proven diagnosis of prostate adenocarcinoma diagnosed by prostate biopsy with archival biopsy tissue available for analysis. The amount of cancer tissue present must be sufficient for analysis.
5. Prostate adenocarcinoma classified as intermediate or high-risk as defined by one or more of the following criteria: PSA >10 ng/ml, Gleason score ≥7, or tumor stage ≥T2b
6. Patients must have no evidence of metastatic disease (including clinically negative pelvic lymph nodes) as established by imaging (CT or MRI of the pelvis and a bone scan) within 60 days prior to registration. Equivocal bone scan findings are allowed if plain film x-rays are negative for metastasis.
7. The patient and the attending urologist have decided to proceed with prostatectomy
8. Lab values meeting the following criteria

   1. Total bilirubin < 2.0 X Upper Limit of Normal (ULN)
   2. Aspartate aminotransferase (AST) ≤ 2.5 X ULN.
   3. Alanine aminotransferase (ALT ) ≤ 2.5 X ULN
   4. Absolute Neutrophil Count (ANC) > 1.5 K/mm3
   5. Platelets > 100 K/mm3
   6. Hemoglobin ≥9.0 g/dL
   7. calculated creatinine clearance ≥ 40 mL/min

   Exclusion Criteria:
9. Patients with low risk prostate adenocarcinoma as defined by meeting all three of the following criteria: Gleason score ≤6, PSA <10 and tumor stage ≤T2b
10. The presence of metastatic disease including to pelvic lymph nodes
11. Use of any beta-blocker at the time of diagnostic biopsy for prostate cancer or use of any beta-blocker at the time of screening. If the investigator does not believe that carvedilol can be safely added to the patients existing antihypertensive regimen, then the patient is not eligible for this study.
12. Prior therapy for prostate cancer including radiation therapy (external beam or brachytherapy), surgery, high-intensity focused ultrasound (HIFU), cryotherapy, previous hormonal therapy with androgen deprivation therapy by bilateral orchiectomy or LHRH analogues (e.g. leuprolide, goserelin, triptorelin, degarelix), antiandrogens, ketoconazole, abiraterone or chemotherapy (for prostate cancer, chemotherapy in the past for other indications is allowed).
13. Treatment with any investigational agent within 30 days prior to being registered for protocol therapy.
14. No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least 5 years.
15. Inability to take oral medication
16. Hypotension (systolic blood pressure <100 mm Hg or diastolic blood pressure <50 mm Hg) or bradycardia (pulse <55 beats/min) at screening. For patients with a functioning pacemaker, bradycardia is not an exclusion.
17. Bronchial asthma or related bronchospastic conditions such as chronic obstructive pulmonary disease.
18. Patients must not have New York Heart Association Class III or IV heart failure at the time of screening. Patients must not have any unstable angina, myocardial infarction, or serious uncontrolled cardiac arrhythmia within 6 months prior to registration.
19. Prolonged QTc interval on pre-entry 12-lead ECG (> 460 msec), obtained within 28 days prior to being registered on study. No second- or third-degree atrioventricular block on screening 12-lead ECG.
20. Any other serious illness or medical condition that the principal investigator feels would make the patient a poor candidate for this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Biomarkers in Prostate Biopsy Compared to Prostatectomy Tissues | 28 days after beginning carvedilol
  BIomarker

SECONDARY OUTCOMES:
Change in Serum PSA | 28 days after beginning carvedilol
  PSA

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magnon C, Hall SJ, Lin J, Xue X, Gerber L, Freedland SJ, Frenette PS. Autonomic nerve development contributes to prostate cancer progression. Science. 2013 Jul 12;341(6142):1236361. doi: 10.1126/science.1236361. PMID 23846904